CLINICAL TRIAL: NCT02368470
Title: Randomized Study on Efficacy of Gemifloxacin-based Regimen for Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyuk Lee, Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2014-07-146-001
Record Dates: First submitted 2015-02-09; First posted 2015-02-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Gemifloxacin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard triple therapy (Active Comparator): Rabeprazole (Rabiet®, ildong pharmaceutical Co. Ltd., Seoul, Korea) 20 mg twice daily, amoxicillin (Pamoxin®, Dongwha Co. Ltd., Seoul, Korea) 1 g twice daily, and clarithromycin (Klaricid®, Abbot Korea Co. Ltd., Seoul, Korea) 500 mg twice daily for 7 days
  Interventions: Drug: Standard triple therapy
- Gemifloxacin-based triple therapy (Experimental): Rabeprazole (Rabiet®, ildong pharmaceutical Co. Ltd., Seoul, Korea) 20 mg twice daily, amoxicillin (Pamoxin®, Dongwha Co. Ltd., Seoul, Korea) 1 g twice daily, and gemifloxacin (Factive®, LG Life Sciences, Ltd, Seoul, Korea) 320 mg once daily for 7 days
  Interventions: Drug: Gemifloxacin-based triple therapy

INTERVENTIONS:
Drug: Gemifloxacin-based triple therapy — Rabeprazole (Rabiet®, ildong pharmaceutical Co. Ltd., Seoul, Korea) 20 mg twice daily, amoxicillin (Pamoxin®, Dongwha Co. Ltd., Seoul, Korea) 1 g twice daily, and gemifloxacin (Factive®, LG Life Sciences, Ltd, Seoul, Korea) 320 mg once daily for 7 days
  Other Names: Factive, Rabiet, Pamoxin
  Arms: Gemifloxacin-based triple therapy
Drug: Standard triple therapy — Rabeprazole (Rabiet®, ildong pharmaceutical Co. Ltd., Seoul, Korea) 20 mg twice daily, amoxicillin (Pamoxin®, Dongwha Co. Ltd., Seoul, Korea) 1 g twice daily, and clarithromycin (Klaricid®, Abbot Korea Co. Ltd., Seoul, Korea) 500 mg twice daily for 7 days
  Other Names: Klaricid, Rabiet, Pamoxin
  Arms: Standard triple therapy

SUMMARY:
New generations of fluoroquinolones, like levofloxacin and moxifloxacin, exhibit a broad-spectrum activity against Gram-positive and Gram-negative bacteria, and have been successfully introduced into the treatment of Helicobacter pylori infection. However, it was suggested that resistance to fluoroquinolones has been increasing in the Korean population and the resistance is most likely mediated through point mutation in gyrA. Gemifloxacin (FACTIVE®) is an enhanced-affinity, broad-spectrum fluoroquinolone suitable for once-daily, oral dosing. In vitro studies have shown that gemifloxacin displays potent activity against Gram-positive organisms, whilst retaining good activity against Gram-negative organisms. Gemifloxacin is the most potent member of the quinolone class against S. pneumoniae with activities 16-64 times greater than those of ciprofloxacin and ofloxacin and 2-8 times greater than those of moxifloxacin. Importantly, gemifloxacin displays potent in vitro activity against strains of S. pneumoniae with known resistance to β-lactams, macrolides and other members of the quinolone class. This potent activity is believed to be due to the enhanced affinity of gemifloxacin for topoisomerase IV, the major fluoroquinolone target in S. pneumoniae. Furthermore, gemifloxacin displays potent activity against H. influenzae and M. catarrhalis and atypical organisms such as L. pneumophila, C. pneumoniae and M. pneumoniae. It has proven particularly effective in respiratory and urinary tract infection.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and the safety of using standard triple therapy and gemifloxacin-containing triple therapy as a first-line treatment for Helicobacter pylori eradication in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-70 years with H. pylori infection
* The presence of H. pylori was defined as positive if the results of one of the following two tests were positive:

  1. Rapid urease test (CLO™, Delta West, Bentley, Western Austria)
  2. Histology. Biopsy specimens, obtained by endoscopy, were fixed in formalin and used for determination of H. pylori infection by Giemsa staining.

Exclusion Criteria:

1. Patients with previous H. pylori eradication therapy
2. Patients treated with H2 receptor antagonist, PPI, and antibiotics in the previous 4 weeks, or nonsteroidal anti-inflammatory drug (NSAID) in the previous 2 weeks
3. Pregnant or lactating women
4. Patients who suffered from serious diseases such as severe liver disease, renal disease, and cerebrovascular disease
5. Patients who had a drug allergy to the study drugs
6. Patients with previous gastric surgery.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk Lee, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea